CLINICAL TRIAL: NCT06118281
Title: ARTEMIS - Effects of Ziltivekimab Versus Placebo on Cardiovascular Outcomes in Patients With Acute Myocardial Infarction
Brief Title: ARTEMIS - A Research Study to Look at How Ziltivekimab Works Compared to Placebo in People With a Heart Attack
Acronym: ARTEMIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX6018-4979; U1111-1294-3473 (Other: World Health Organization (WHO)); 2023-506876-28 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Risk; Acute Myocardial Infarction (AMI)
MeSH Terms: interventions — ziltivekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ziltivekimab (Experimental): Participants will receive an initial loading dose of ziltivekimab Dose 1 subcutaneously (s.c.) as early as possible after invasive procedure, and latest within 36 hours of hospitalisation for ST-elevation myocardial infarction (STEMI) and within 48 hours of hospitalisation for non-ST-elevation myocardial infarction (NSTEMI), followed by ziltivekimab Dose 2 s.c. once-monthly during the treatment period (estimated up to 2 years) added to standard of care.
  Interventions: Drug: Ziltivekimab
- Placebo ziltivekimab (Experimental): Participants will receive placebo matched to ziltivekimab at an initial loading dose subcutaneously (s.c.) as early as possible after invasive procedure, and latest within 36 hours of hospitalisation for STEMI and latest within 48 hours of hospitalisation for NSTEMI, followed by placebo matched to ziltivekimab s.c. once-monthly during the treatment period (estimated up to 2 years) added to standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziltivekimab — Ziltivekimab will be adminsitered subcutaneously as an initial loading dose of Dose 1 followed by a maintenance dose of Dose 2 once- monthly.
  Arms: Ziltivekimab
Drug: Placebo — Placebo matched to ziltivekimab will be adminsitered subcutaneously as an initial loading dose followed by a maintenance dose once-monthly.
  Arms: Placebo ziltivekimab

SUMMARY:
The research study is being done to see if ziltivekimab can be used to treat people who were admitted to hospital because of a heart attack. Ziltivekimab might reduce development of heart disease, thereby preventing new heart attacks or strokes. Participants will either get ziltivekimab (active medicine) or placebo (a dummy medicine which has no effect on the body). Which treatment participants get is decided by chance. The chance of getting ziltivekimab or placebo is the same. The participant will need to inject the study medicine into a flat skin surface in there stomach, thigh, or upper arm once every month. Ziltivekimab is not yet approved in any country or region in the world. It is a new medicine that doctors cannot prescribe. The study will last for about 2 years.

ELIGIBILITY:
Key inclusion:

* Age 18 years or above at the time of signing the informed consent.
* Hospitalisation for acute myocardial infarction with evidence of type 1 myocardial infarction (MI) by invasive angiography performed at site with percutaneous coronary intervention (PCI) capabilities.
* ST-segment elevation myocardial infarction (STEMI) with all the following: a) Relevant onset of symptoms suggestive of cardiac ischaemia within 12 hours before hospitalisation, at the investigator's discretion.

  b) Electrocardiogram (ECG)-changes (in the absence of left ventricular hypertrophy or left bundle branch block): ST-segment elevation at the J point in at least two contiguous leads greater than or equal 0.25 (millivolt) mV in men less than 40 years, greater than or equal 0.2 mV in men greater than or equal 40 years, or greater than or equal 0.15 mV in women in leads V2-V3; and/or greater than or equal 0.1 mV in all other leads.

OR

* Non-ST-segment myocardial infarction with all the following: a) Relevant onset of symptoms suggestive of cardiac ischaemia within 24 hours before hospitalisation, at the investigator's discretion. b) Rise and/or fall in car-diac troponin I or T with at least one value above the 99th percentile upper reference limit.
* Possibility for both randomisation and administration of the loading dose of study intervention as early as possible after invasive procedure, and latest within 36 hours of hospitalisation (time 0) for STEMI, and latest within 72 hours of hospitalisation (time 0) for NSTEMI.
* Presence of at least one of the following criteria confirmed based on the participant's medical records and/or medical history interview: a) Any prior MI. b) Prior coronary revascularisation. c) Diabetes mellitus treated with ongoing glucose-lowering agent(s). d)Known chronic kidney disease (CKD) (estimated glomerular filtration rate (eGFR) greater than or equal to 15 and less than 60 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2). e) Prior ischaemic stroke. f) Known carotid disease or peripheral artery disease in the lower extremities. g) Multivessel coronary artery disease (current/prior). h) For STEMI patients only: anterior MI at index acute myocardial infarction (AMI)

Key exclusion:

* Use of fibrinolytic therapy for treatment of the current AMI.
* Chronic heart failure classified as being in New York Heart Association (NYHA) Class IV.
* Ongoing haemodynamic instability defined as any of the following: a) Killip Class III or IV. b) Sustained and/or symptomatic hypotension (systolic blood pressure less than 90 millimeters of mercury (mmHg)).
* Severe kidney impairment defined as any of the following: a) eGFR less than 15 mililitre per minute per 1.73 m^2. b) Chronic haemodialysis or peritoneal dialysis.
* Known alanine aminotransferase (ALT) greater than 8 x upper limit of normal (reference range) (ULN).
* Severe hepatic disease defined as at least one of the following: a) Previously known or current hepatic encephalopathy (clinical evaluation). b) Previously known or current ascites (clinical eval-uation). c) Jaundice (clinical evaluation). d) Previous oesophageal/gastric variceal bleeding. c) Known hepatic cirrhosis.
* Major cardiac surgical (including but not restricted to coronary artery bypass graft surgery (CABG)), non-cardiac surgical, or major endoscopic procedure (thoracoscopic or laparoscopic) within the past 60 days or any major surgical procedure planned at the time of randomisation or as treatment for the current AMI (CABG). Deferred (staged)percutaneous coronary intervention for a non-culprit vessel identified during the current AMI is allowed.
* Clinical evidence of, or suspicion of, active infection at the discretion of the investigator.
* Known (acute or chronic) hepatitis B or hepatitis C.
* History or evidence of untreated latent tuberculosis (TB) such as (but not limited to): a) History of a positive TB test or chest X-ray compatible with latent TB; and TB treatment initiated less than 28 days prior to randomisation. b) Participants with TB risk factors but unwilling to undergo TB treatment if confirmed positive for latent TB based on central laboratory test at baseline (visit 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of a 3-component major adverse cardiovascular event (MACE) endpoint comprising: Cardiovascular (CV) death, Non-fatal myocardial infarction (MI), Non-fatal stroke | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.

SECONDARY OUTCOMES:
Number of CV death, non-fatal MI, non-fatal stroke | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as count of events.
Time to first occurrence of a composite MACE endpoint consisting of: All-cause mortality, Non-fatal MI, Non-fatal stroke | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Number of all-cause mortality, non-fatal MI, non-fatal stroke | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as count of events.
Time to first occurrence of non-fatal MI | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Time to first occurrence of MI (fatal and non-fatal) | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Time to first occurrence of non-fatal stroke | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Time to first occurrence of stroke (fatal and non-fatal) | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Time to first occurrence of a 3-component coronary MACE endpoint comprising:CV death, Non-fatal MI, Ischaemia-driven coronary revascularisation | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Time to first occurrence of a 5-component expanded MACE endpoint comprising: CV death, Non-fatal MI, Non-fatal stroke, Ischaemia-driven coronary revascularisation, Heart failure (HF) hospitalisation or urgent HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Number of CV death, non-fatal MI, non-fatal stroke, ischaemia-driven coronary revascularisation, or HF hospitalisation or urgent HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measired as count of events.
Time to first occurrence of a 3-component HF endpoint comprising: CV death, HF hospitalisation or urgent HF visit, Outpatient HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Number of CV deaths, HF hospitalisation or urgent HF visits or outpatient HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in count of events.
Time to first occurrence of a 2-component HF endpoint comprising: CV death, HF hospitalisation or urgent HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as months.
Number of CV deaths, HF hospitalisation or urgent HF visits | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in count of events.
Time to first occurrence of a 2-component expanded HF endpoint comprising: HF hospitalisation or urgent HF visit, Outpatient HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as months.
Number of HF hospitalisation or urgent HF visit or outpatient HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as count of events.
Number of outpatient HF visit | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in count of events.
Time to occurrence of CV death | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as months.
Time to occurrence of all-cause death | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as months.
Time to first occurrence of 6-component vascular event endpoint: CV death, Non-fatal MI, Non-fatal stroke, Ischaemia-driven coronary revascularisation, Non-coronary revascularisation procedure, Any other non-coronary ischaemic event excluding stroke | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Number of CV death, non-fatal MI and non-fatal stroke, ischaemia-driven coronary revascularisation, non-coronary revascularisation procedure, or any other non-coronary ischaemic event excluding stroke | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as count of events.
Number of ischaemia-driven coronary revascularisation | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as count of events.
Time to first occurrence of ischaemia-driven coronary revascularisation or any non-coronary revascularisation | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured in months.
Number of ischaemia-driven coronary revascularisation or any non-coronary revascularisation | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as count of events.
Number of cardiovascular hospitalisations | From randomisation (month 0) to 1 month/ 30 days
  Measured as count of events.
Number of cardiovascular hospitalisations | From randomisation (month 0) to 12 months
  Measured as count of events.
Number of hospitalisations with infection as primary cause or death due to infection | From randomisation (month 0) to end-of-study (up to 25 months)
  Measured as count of events.
Change in high-sensitivity C-reactive protein (hs-CRP) | From randomisation (month 0) to 6 months
  Measured as ratio to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (823):
- United States (188):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Grandview Medical Center, Birmingham, Alabama
  - Eastern Shore Rsrch Inst, LLC, Fairhope, Alabama
  - Heart Center Rsrch_Hunstville, Huntsville, Alabama
  - Mobile Heart USA Health Cardiology Clinic, Mobile, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - Arkansas Cardiology Clinic, Little Rock, Arkansas
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Valley Clinical Trials, Covina, California
  - UCSD Medical Center, La Jolla, California
  - Loma Linda University Faculty Medical Clinics, Loma Linda, California
  - VAGrtrLosAngelesHlthcareSystem, Los Angeles, California
  - University of Californ LA-UCLA, Los Angeles, California
  - University Of California Irvine, Orange, California
  - Kaiser Permanente Viewridge Medical Offices, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - San Francisco V.A. Medical Center, San Francisco, California
  - LA BioMed Harbor UCLA Med Cenr, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Interventional Cardiology Medical Group, West Hills, California
  - University of CO - Division of Cardiology, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Colorado Heart and Vascular PC, Golden, Colorado
  - S Denver Cardiology Associates, Littleton, Colorado
  - Advanced Heart & Vein Center, Thornton, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Danbury Hospital - Cardiology Department, Danbury, Connecticut
  - Yale Ctr for Clin Invest, New Haven, Connecticut
  - Cardiology Associates of Fairfield County, Stamford, Connecticut
  - Christiana Care Health Services, Inc., Newark, Delaware
  - MedStar Hlth Res Institute, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Healthcare, Hollywood, Florida
  - UF Hlth Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Baptist Heart Specialists, Jacksonville, Florida
  - Baptist Hospital Cardiology, Pensacola, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Atlanta VAMC, Decatur, Georgia
  - Northeast Georgia Medical Ctr, Gainesville, Georgia
  - Cardio. Consult. of S. GA, Thomasville, Georgia
  - St. Luke's Idaho Cardiology Associates, Meridian, Idaho
  - Endeavor Health Glenbook Hosp, Evanston, Illinois
  - OSF HealthCare_Cardiovasc Inst, Rockford, Illinois
  - Prairie Cardiovascular Consultants, Ltd., Springfield, Illinois
  - Midwest Cardiovascu Rsrch Foundation, Elkhart, Indiana
  - Indiana University Health Methodist Hosptial, Indianapolis, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - MercyOne NE Iowa Fam Med & Res, Waterloo, Iowa
  - University Of Kansas Hospital, Kansas City, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Saint Elizabeth Medical Center, Edgewood, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Overton Brooks V.A. Medical Center, Shreveport, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center Bramhall, Portland, Maine
  - MedStar Hlth Res Institute, Clinton, Maryland
  - Adventist HealthCare Shady Grove Medical Center, Rockville, Maryland
  - Jadestone Clinical Research, LLC, Silver Spring, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - McLaren Bay Region, Bay City, Michigan
  - Wayne State University/University Health Center, Detroit, Michigan
  - WMU Homer Stryker MD School of Medicine, Kalamazoo, Michigan
  - McLaren Greater Lansing, Lansing, Michigan
  - MidMic Medical Cntr - Midland, Midland, Michigan
  - McLaren Macomb Health Care, Mount Clemens, Michigan
  - McLaren Northern MI Hosp, Petoskey, Michigan
  - Trinity Health Oakland Hospital, Pontiac, Michigan
  - Corewell Health, Royal Oak, Michigan
  - Ascension St. Mary's Research Institute - Michigan, Southfield, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Essentia Health, Duluth, Minnesota
  - Fairview Health Services, Maplewood, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - VA Medical Center_Minneapolis, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Univ of Mississippi Med Center, Jackson, Mississippi
  - Cardiolg Assoc Rsch LLC_Tupelo, Tupelo, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Missouri Cardiovascular Specialist, Columbia, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Research, Springfield, Missouri
  - Washington University School of Medicine_St. Louis, St Louis, Missouri
  - Methodist Physicians Clinic, Omaha, Nebraska
  - UMC of Southern Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Med Ctr, Lebanon, New Hampshire
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Virtua Health, Camden, New Jersey
  - Hackensack Meridian Health, Hackensack, New Jersey
  - The Heart House Haddon Heights, Haddon Heights, New Jersey
  - Jersey City Med Center, Jersey City, New Jersey
  - Inspira Health, Mullica Hill, New Jersey
  - AtlantiCare Regional Medi Cnt, Pomona, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Vineland, New Jersey
  - The New York Hospital, Brooklyn, New York
  - Trinity Medical WNY, PC, Buffalo, New York
  - Saint Joseph's Hospital Health Center, Liverpool, New York
  - NYU Grossman School of Med, New York, New York
  - Mount Sinai Morningside, New York, New York
  - University of Rochester, Rochester, New York
  - St Francis Hospital Lindner Research Center, Roslyn, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Jacobi Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Cardiology Associates_Asheville, Asheville, North Carolina
  - UNC Hospital HVC_Meadowmont, Chapel Hill, North Carolina
  - Novant Hlth Vasc Ins Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moses H. Cone Mem Hosp, Greensboro, North Carolina
  - Wake Forest Uni Hlth Sciences, High Point, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Novant Hlth Cardio - Kimel Park, Winston-Salem, North Carolina
  - Sanford Health - Fargo, Fargo, North Dakota
  - Trinity Medical Group, Minot, North Dakota
  - Aultman Hospital, Canton, Ohio
  - Lindner Center,Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati/UC Health, Cincinnati, Ohio
  - Louis Stokes Clvlnd VA Med Ctr, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic_Cleveland, Cleveland, Ohio
  - University Hospitals Of Cleveland Medical Center, Elyria, Ohio
  - Wright State University, Fairborn, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - ProMedica, Toledo, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Genesis Health Care System, Zanesville, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Penn State Hlth Holy Spirit Med Ctr, Camp Hill, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health Clinical Research, Anderson, South Carolina
  - Prism Hlth Carolina Card Cons, Greenville, South Carolina
  - Monument Health Clinical Rsrch, Rapid City, South Dakota
  - Sanford Research, Sioux Falls, South Dakota
  - Chattanooga Heart Institute, Chattanooga, Tennessee
  - Knoxville Heart Group, Knoxville, Tennessee
  - Tennova HC Turkey Creek MC, Knoxville, Tennessee
  - Baptist Clin Res Institute, Memphis, Tennessee
  - Saint Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Parkway Cardiology Associates, PC, Oak Ridge, Tennessee
  - CV Research of Knoxville, Powell, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Austin Heart, Austin, Texas
  - Liver Ins@ Mthdist DTX Med Cen, Dallas, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Heart Inst Medical Ctr, Houston, Texas
  - UT Health University of Texas, Houston, Texas
  - Prolato Clinical Research Cntr, Houston, Texas
  - HCA Research Institute, McAllen, Texas
  - Heart & Vascular Inst._Titus, Mount Pleasant, Texas
  - Baylor Scott & White Res Inst, Plano, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Christus Heart and Vascular Institute, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Sentara Bayside Hospital, Norfolk, Virginia
  - Chippenham Medical Center, Richmond, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, LLC, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - VA Medical Center_Salem, Salem, Virginia
  - Valley Health Link, Winchester, Virginia
  - Swedish Medical Center_Seattle, Seattle, Washington
  - University Of Washington_Seattle, Seattle, Washington
  - Multicare Health System, Tacoma, Washington
  - Aurora St. Luke's Medi Ctr, Milwaukee, Wisconsin
- Argentina (19):
  - Instituto Cardiovascular Buenos Aires, CABA, Buenos Aires
  - Hospital Italiano de la Plata, La Plata, Buenos Aires
  - Hospital Universitario Austral - Instituto de Cardiologia, Pilar, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Sanatorio Modelo Quilmes, Quilmes, Buenos Aires
  - Fundación Nuestra Señora del Rosario - Estudios Clínicos los Arroyos, San Nicolás de los Arroyos, Buenos Aires
  - Fundacion Favaloro, CABA, Buenos Aires, Argentina
  - Sanatorio Güemes, CABA, City of Buenos Aires
  - Hospital Español de Mendoza, Godoy Cruz, Mendoza, Mendoza Province
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Hospital del Centenario, Rosario, Santa Fe, Santa Fe Province
  - Centro Privado de Cardiología, San Miguel de Tucuimán, Tucumán Province
  - Centro de Investigación C.I.C.E 9 de Julio - Sanatorio 9 de Julio, San Miguel de Tucumán, Tucumán Province
  - Sanatorio Finochietto, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Cardiología Hospital J. M. Ramos Mejia, Buenos Aires
  - Instituto de Cardiología de Corrientes, Corrientes
  - Clínica Privada Velez Sarsfield, Córdoba
  - Hospital Dr. Jose Maria Cullen, Santa Fe
- Australia (23):
  - Concord Repatriation General Hospital - Cardiology Department, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital_Randwick, Randwick, New South Wales
  - Illawarra Heart Health Centre, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Brisbane, Queensland
  - Cairns Base Hospital, Cairns, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Gold Coast University Hospital - Cardiology Department, Southport, Queensland
  - Gold Coast University Hosptial, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital Cardiovascular Clinical Trials, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Northern Health, Epping, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Adrian Costa Clinical Trials Centre, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, South Yarra, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Brazil (22):
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Hospital Ruy Azeredo Ltda, Goiânia, Goiás
  - NUPEC Cardio, Belo Horizonte, Minas Gerais
  - Irmandade Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital Maternidade e Pronto Socorro Santa Lúcia, Poços de Caldas, Minas Gerais
  - Hospital das Clínicas da Universidade Federal do Triangulo Mineiro, Uberaba, Minas Gerais
  - Centro de Pesquisa Clínica do Hospital de Clínicas da Universidade Federal de Uberlândia, Uberlândia, Minas Gerais
  - Hospital Agamenon Magalhães, Recife, Pernambuco
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas - PUC/RS, Porto Alegre, Rio Grande do Sul
  - Associação Lar São Francisco de Assis na Providência de Deus - Bragança Paulista, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - PUCCAMP - Hospital e Maternidade Celso Pierro, Campinas, São Paulo
  - Integral Pesquisa e Ensino, Cidade Nova Votuporanga, São Paulo
  - Irmandade da Santa Casa de Misericórdia de Marília, Marília, São Paulo
  - Hospital Israelita Albert Einstein, Morumbi, São Paulo
  - ASSOCIAÇÃO LAR SÃO FRANCISCO DE ASSIS NA PROVIDÊNCIA DE DEUS - Hospital Regional de Presidente Prudente, Presidente Prudente, São Paulo
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
  - Jmf Clínica Do Coração Ltda, Aracaju
  - Hospital Mãe de Deus - Porto Alegre, Porto Alegre/RS
- Bulgaria (34):
  - MHAT "Puls" AD Cardiology Department, Blagoevgrad
  - MHAT Heart and Brain EAD, Burgas
  - UMHAT - Burgas AD, Burgas
  - UMHAT Deva Maria EOOD, Burgas
  - MHAT Dr. Tota Venkova AD, Gabrovo
  - Multiprofile Hospital For Active Treatment Dr. Tota Venkova AD, Gabrovo
  - MHAT - Ivan Skenderov EOOD, Gotse Delchev
  - MHAT Haskovo AD, Haskovo
  - MHAT - Dr. Atanas Dafovski AD, Cardiology department, Kardzhali
  - MHAT - Cardiolife OOD - Lovech, Lovech
  - MHAT - City Clinic - Sveti Georgi EOOD, Montana
  - "MHAT - Pazardzhik", Pazardzhik
  - MHAT Heart and Brain, Pleven
  - UMHAT Pulmed, Department of Cardiology, Plovdiv
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Cardiology, Plovdiv
  - MHAT MC-Sv Ivan Rilski EOOD, Plovdiv
  - MHAT Sveta Karidad EAD, Plovdiv
  - SHATC - Medica Kor EAD, Rousse
  - MHAT Southwest Hospital OOD, Cardiology Department, Sandanski
  - MHAT Hadzhi Dimitar OOD, Sliven
  - MHAT "Dr. Bratan Shukerov", Smolyan
  - MHAT Dr. Bratan Shukerov, Smolyan
  - Mhat "Nch", Sofia
  - Acibadem City Clinic UMHAT Tokuda EAD, Cardiology, Sofia
  - Acibadem City Clinic UMHAT EOOD, Cardiology, Sofia
  - "UMHAT "Aleksandrovska" EAD, Cardiology clinic, Sofia
  - UMHAT Sveta Ekaterina EAD, Sofia
  - UMHATEM N.I. Pirogov EAD, Sofia
  - "UMHAT "Sveta Anna" Sofia" AD, Clinic of Cardiology, Sofia
  - UMHAT Sofiamed EAD, Sofia
  - SHATC - Cardiolife OOD - Varna, Varna
  - Specialized Hospital For Active Cardiology Treatement Cardiolife OOD, Varna
  - UMHAT "Sveta Marina" EAD, Varna
  - SHATC - Yambol EAD, Yambol
- Canada (32):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Univ of Alberta Hosp Edmonton, Edmonton, Alberta
  - Kelowna Cardiology Res. Ltd., Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint Paul's Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - New Brunswick Heart Centre, Saint John, New Brunswick
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Hel Bra Civic Hs, Brampton, Ontario
  - Health Sciences North Rsrch Inst, Greater Sudbury, Ontario
  - Hamilton Health Sciences Corp, Ontario, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Center Ontario, London, Ontario
  - Southlake Regional Hlth Centre, Newmarket, Ontario
  - University of Ottawa Heart Ins, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - UHN-Toronto General Hospital, Toronto, Ontario
  - CIUSS Hopit de Chicoutimi, Chicoutimi, Quebec
  - CHUM Centre de Recherch Hotel-Dieu, Montreal, Quebec
  - Hopital Sacre-Coeur de Montreal, Montreal, Quebec
  - CISSS de Lanaudiere - Centre hospitalier De Lanaudiere, Saint-Charles-Borromée, Quebec
  - CISSSL Hôsp Pierre-Le Gardeur, Terrebonne, Quebec
  - Centre hosp affilié univ rég, Trois-Rivières, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
  - CHU de Quebec-Universite-Laval,HDQ, Québec
  - Ins Uni de Cardi et de PNA de, Québec
- China (45):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital-Cardiology, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology-Cardiology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University-Cardiology, Wuhan, Hubei
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - China-Japan Union Hospital of Jilin University-Cardiology, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The People's Hospital of Liaoning Province-Cardiology, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University-Cardiology, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an JiaoTong University-Cardiovascular, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Zhongshan Hospital, Fudan University-Cardiology, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University-Cardiology, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital-Cardiology, Chengdu, Sichuan
  - General Hospital of Tianjin Medical University-Endocrinology, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - TEDA International Cardiovascular Hospital-Cardiovascular, Tianjin, Tianjin Municipality
  - TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital-Cardiology, Hangzhou, Zhejiang
  - The 1st Affiliated Hospital of WMU-Cardiology, Wenzhou, Zhejiang
  - The First Affiliated Hospital of WMU-Cardiology, Wenzhou, Zhejiang
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Zhongda Hospital, Southeast University, Nanjing
  - Shengjing Hospital of China Medical University, Shenyang
- Czechia (14):
  - Krajská nemocice Liberec, a.s, Liberec, Czech Republic
  - Krajská zdravotní, a.s. - Masarykova nemocnice v Ústí nad Labem, o.z., Ústní Nad Labem, Czechia
  - Fakultni nemocnice Brno, Brno
  - FN u Sv. Anny, Brno
  - Nemocnice České Budějovice a.s., České Budějovice
  - Fakultní nemocnice Olomouc, Olomouc
  - Nemocnice Pardubickeho kraje a.s., Pardubice
  - Fakultni nemocnice Plzen - Lochotin, Plzen - Lochotín
  - Fakultní nemocnice Královské Vinohrady, Prague
  - II. interni klinika VFN - Kardiologie a angiologie, Prague
  - IKEM, Prague
  - Nemocnice na Homolce, Prague
  - Nemocnice AGEL Třinec-Podlesí a.s., Třinec
  - Krajská nemocnice T.Bati a.s., Zlín
- Denmark (7):
  - Herlev og Gentofte Hospital, Hellerup, Capital Region
  - Aalborg Universitetshospital Kardiologisk Afdeling, Aalborg
  - Aarhus Universitetshospital, Hjertesygdomme, Aarhus N
  - Nordsjællands hospital - Kardiologisk Forskning, Hillerød
  - Rigshospitalet - Kardiologisk Forskningsenhed, København Ø
  - Odense Universitetshospital, Kardiologisk afd., Odense C
  - Svendborg Sygehus - Kardiologisk, Svendborg
- France (19):
  - Centre Hospitalier Universitaire de Besancon-Hopital Jean Minjoz, Besançon
  - Hospices Civils de Lyon- Hopital Louis Pradel, Bron
  - Centre Hospitalier Universitaire de Caen Normandie- Cote de Nacre, Caen
  - Centre Hospitalier Regional Universitaire de Tours-Hopital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon, Grenoble
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier Universitaire de Lille-Institut Coeur Poumon, Lille
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Assistance Publique Hopitaux de Marseille-Hopital de La Timone-1, Marseille
  - Centre Hospitalier Universitaire de Nice-Hopital Pasteur, Nice
  - Aphp-Hopital La Pitie Salpetriere-1, Paris
  - Ap-Hp-Hopital Europeen Georges Pompidou, Paris
  - Ap-Hp-Hopital Bichat-Claude Bernard-1, Paris
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-1, Toulouse
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil, Toulouse
  - Chru de Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (28):
  - Rhön-Klinikum AG - Zentralklinik Bad Berka - Kardiologie, Bad Berka
  - Charité - Campus Benjamin Franklin - Klinik für Kardiologie, Berlin
  - BG Klinikum Unfallkrankenhaus Berlin GmbH - Klinik für Kardiologie, Berlin
  - Uniklinik Klinikum Bielefeld - Kardiologie und Internist. Intensivmedizin, Bielefeld
  - Bremer Institut für Herz- und Kreislaufforschung (BIHKF), Bremen
  - Cellitinnen-Krankenhaus St. Vinzenz Köln - Kardiologie, Cologne
  - Amper Kliniken AG - Helios Amper-Klinikum Dachau - Kardiologie, Dachau
  - Kath. St. Paulus GmbH - St Johannes Hospital Dortmund - Kardiologie, Dortmund
  - Städt. Klinikum Dresden - 2. Medizinische Klinik, Dresden
  - Uniklinik TU Dresden - Herzzentrum Dresden GmbH, Dresden
  - Universitätsklinikum Düsseldorf - Klinik für Kardiologie, Pneumologie und Angiologie, Düsseldorf
  - Helios Klinikum Erfurt GmbH - 3. Med. Klinik - Kardiologie, Erfurt
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Universitätsklinikum Frankfurt aM - Kardiologie, Frankfurt am Main
  - Universitätsklinikum Freiburg - Medical Center, Freiburg im Breisgau
  - Klinikum Friedrichshafen GmbH - Klinik für Kardiologie, Angiologie, Pneumologie und internistische Intensivmedizin, Friedrichshafen
  - Klinikum Fulda gAG - Med. Klinik I, Fulda
  - Universitätsklinikum Hamburg-Eppendorf - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover - Kardiologie und Angiologie, Hanover
  - UniklinikHeidelberg - Innere Med. III - Kardiologie, Angiologie, Pneumologie, Heidelberg
  - Asklepios Klinik Langen - Medizinische Klinik I, Langen
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Kardiologie, Leipzig
  - Klinikum Leverkusen gGmbH - Med. Klinik 1, Leverkusen
  - Universitätsklinikum Mannheim - 1. Medizinische Klinik, Mannheim
  - Deutsches Herzzentrum TU München - Klinik für Herz- und Kreislauferkrankungen, München
  - Uniklinik Regensburg - Innere Medizin II, Regensburg
  - Robert-Bosch-Krankenhaus GmbH Stuttgart, Stuttgart
  - Uniklinik Tübingen - Innere Med. III Kardiologie und Angiologie, Tübingen
- Greece (31):
  - Univ Gen Hospital Larisa, Cardiology Medicine Clinic, Larissa/Thessaly, Greece
  - General Hospital Of Thessaloniki Papageorgiou, Nea Efkarpia, Thessaloniki
  - General Hospital of Athens "Elpis", Ampelokipoi/Athens
  - Evangelismos Hospital, Athens
  - G.H. of Athens "Evaggelismos", Athens
  - NIMTS Army Share Fund Hospital, Athens
  - Group Euroclinic - Athens Euroclinic, Athens
  - Henry Dunant Hospital Center, Athens
  - "Sotiria" Thoracic Diseases Hospital of Athens, Athens
  - 'G. Gennimatas' General Hospital of Athens, Athens
  - Hippokration Hospital, Athens
  - Thoracic General Hospital Of Athens I Sotiria - Cardiology Department, Athens
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - Konstantopouleio G.H. of Athens, "Agia Olga", Athens
  - "Hygeia" General Hospital of Athens, Athens
  - Metropolitan General Hospital Healthcare Facilities Operation And Management Single Member S.A. - Cardiology Clinic, Athens
  - Asklepieion General Hospital - Cardiology Clinic, Athens/Voula
  - U.G.H of Athens "Attikon", Chaidari, Athens
  - General Hospital of Chios "Skilitsio" - Cardiology Clinic, Chios
  - General Hospital Of Eleusina Thriasio - Cardiology Clinic, Eleusina
  - General Hospital of Athens "LAIKO", Goudi/Athens
  - University General Hospital of Ioannina,Internal Medicine, Ioannina
  - Kat Attica General Hospital - Cardiology Clinic, Kifissia
  - Sismanogleio General Hospital - Cardiology Department, Marousi
  - General Hospital Of Patras Agios Andreas - Cardiology Department, Pátrai
  - Geniko Nosokomeio Peiraia Tzaneio - Cardiology department, Piraeus
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - Gen Hospital of Thessaloniki G.Papanikolaou,Cardiology Dpt, Thessaloniki
  - Pan-Arcadian General Hospital of Tripoli Evangelistria - Cardiology Department, Tripoli
  - General Hospital of Imathia Monada Veria, Véroia
- India (58):
  - Lalitha Super Specialities Hospital, Guntur, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Medicover Hospitals, Visakhapatnam MVP, Visakhapatnam, Andhra Pradesh
  - SMC Heart Institute and IVF Research Centre, Raipur, Chhattisgarh
  - Sardar Vallabhbhai Patel Institute of Medical Sciences and Research, Ahmedabad, Gujarat
  - Marengo CIMS Hospital, Ahmedabad, Gujarat
  - Shri B. D. Mehta Mahavir Heart Institute, Surat, Gujarat
  - Sterling Hospitals, Race Course Road, Vadodara, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Ramaiah Memorial Hospital, Bengaluru, Karnataka
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bengaluru, Karnataka
  - Justice K S Hegde Charitable Hospital, Mangaluru, Karnataka
  - Kasturba Medical College and Hospital, Manipal, Udupi, Karnataka
  - Lisie Hospital, Kochi, Kerala
  - Lakshmi Hospital, Palakkad, Kerala
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - Arneja Heart & Multispeciality Hospital, Nagpur, Maharashtra
  - Shri Krishna Hrudayalaya & Critical Care Centre, Nagpur, Maharashtra
  - Central India Cardiology Hospital and Research Institute, Nagpur, Maharashtra
  - All India Institute of Medical Sciences (AIIMS), Nagpur, Nagpur, Maharashtra
  - Chopda Medicare and Research Centre Pvt. Ltd., Nashik, Maharashtra
  - Vijan Hospital & Research Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Atal Bihari Vajpayee Institute of Medical Sciences and Dr. Ram Manohar Lohia Hospital, New Delhi, National Capital Territory of Delhi
  - G B Pant Institute of Postgraduate Medical Education and Research, New Delhi, National Capital Territory of Delhi
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - Fortis Escorts Heart Institute, New Delhi, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - Vardhaman Mahavir Medical College & Safdarjung Hospital, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Batra Hospital and Medical Research Center, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospital, New Delhi, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Bhubaneswar, Odisha
  - SCB Medical College and Hospital, Cuttack, Odisha
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Fortis Hospital, Mohali, Mohali, Punjab
  - S.P. Medical College & Associated Group of Hospitals, Bikaner, Rajasthan
  - SMS Medical College & Attached Hospitals, Jaipur, Rajasthan
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - Sri Ramachandra Medical Centre, Chennai, Tamil Nadu
  - G. Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
  - Jawaharlal Institute of Postgraduate Medical Education and Research (JIPMER), Puducherry, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - ESIC Medical College and Hospital, Hyderabad, Hyderabad, Telangana
  - Malla Reddy Narayana Multispeciality Hospital, Hyderabad, Telangana
  - Jawaharlal Nehru Medical College and Hospital, Aligarh, Uttar Pradesh
  - Ganesh Shankar Vidyarthe Memorial (GSVM) Medical College, Kanpur, Uttar Pradesh
  - King George's Medical University (KGMU), Lucknow, Uttar Pradesh
  - Dr. Ram Manohar Lohia Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
  - B M Birla Heart Research Centre, Kolkata, West Bengal
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - Medical College & Hospital, Kolkata, Kolkata, West Bengal
  - Nil Ratan Sircar Medical College and Hospital, Kolkata, West
  - Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh, Chandigarh
  - Aakash Healthcare Super Speciality Hospital, New Delhi
- Israel (11):
  - Shamir MC - Pediatric and Adolescents Endocrinology unit, Beer Yaakov
  - Hillel Yafe MC - Cardiology Department, Hadera
  - Rambam MC - Cardiac Intensive Care Unit, Haifa
  - Wolfson MC - The Heart Institute, Holon
  - Hadassah Ein Karam MC - Cardio Department, Jerusalem
  - Hadassah Mount Scorpus MC - Cardiology department, Jerusalem
  - Meir MC - Cardiology department, Kfar Saba
  - Rabin MC -Beilinson - Cardiac intensive unit, Petah Tikva
  - Kaplan MC - Cardiac Intensive Care, Rehovot
  - Sourasky MC - Cardio Vascular Research Center, Tel Aviv
  - Sheba MC - Cardiology Clinical Research Unit, Tel Litwinsky
- Italy (40):
  - Ss. Annunziata, Chieti, Abruzzo
  - AORN "Sant'Anna e San Sebastiano", Caserta, Ce
  - A.O.U. Ferrara, Sant'Anna, Cona (Ferrara), Fe
  - ICOT Istituto Marco Pasquali - UOC Cardiologia, Latina, Lazio
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo, Lombardy
  - IRCCS Policlinico San Donato, San Donato Milanese, MI
  - A.O.U Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliera Santa Maria Degli Angeli, Pordenone, PN
  - Azienda Sanitaria Friuli Occidentale - Azienda Ospedaliera Santa Maria Degli Angeli - SC Cardiologia Pordenone, Pordenone, PN
  - Presidio Ospedaliero di Rivoli, Rivoli, To
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano SC Cardiologia, Torino, To
  - Ente Ecclesiastico Ospedale Generale Regionale Miulli - Cardiologia e UTIC, Acquaviva delle Fonti
  - Azienda Ospedaliero-Universitaria SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Maggiore Carlo Alberto Pizzardi, Bologna
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - Ospedale Civile dell'Annunziata, Cosenza
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - AUSL Toscana Sud Est - Ospedale Misericordia Grosseto, Grosseto
  - Ospedale Sant'Andrea - UOC Cardiologia, La Spezia
  - ICOT Istituto Marco Pasquali - UOC Cardiologia, Latina
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - AOU Maggiore della Carità di Novara - Dipartimento Toraco-Cardio-Vascolare - SCDU Cardiologia, Novara
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliera di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Unità Sanitaria Locale Di Piacenza - Cardiologia, Piacenza
  - Arcispedale S Maria Nuova Azienda ULSS-IRCCS, Reggio Emilia
  - AUSL Romagna - Distretto Rimini - Ospedale Infermi, Rimini
  - Ospedale Sandro Pertini - UOC Cardiologia, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Rome
  - Policlinico Casilino - Cardiologia e UTIC, Rome
  - Ospedale Isola Tiberina Gemelli Isola, Rome
  - Azienda Ospedaliero - Universitaria Sant'Andrea, Rome
  - A.O.U Città della Salute e della Scienza di Torino, Torino
  - AOUI Verona, Verona
- Japan (38):
  - Miyazaki Medical Association Hospital_Cardiology, Miyazaki, Miyazaki
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Fujita Health University Hospital_Cardiology, Aichi
  - Toho University Sakura Medical Center_Cardiology, Chiba
  - Asahi General Hospital_Cardiology, Chiba
  - Ehime Prefectural Central Hosp, Ehime
  - Matsuyama Red Cross Hospital_Department of Cardiovascular Medicine, Ehime
  - Japanese Red Cross Fukuoka Hospital_Cardiology, Fukuoka
  - St.Mary's Hospital_Cardiology, Fukuoka
  - Fukuoka University Hospital_Cardiology, Fukuoka-shi, Fukuoka
  - Hyogo Prefectural HarimaHimeji General Medical Center_Cardiology, Himeji-shi, Hyogo
  - Hanaoka Seishu Memorial Hosp._Cardiovascular Medicine, Hokkaido
  - Hanaoka Seishu Memorial Hospital, Hokkaido
  - Nishinomiya Watanabe Cardiovascular Cerebral Center_Cardiovascular Medicine, Hyōgo
  - Hyogo Medical University Hospital_Cardiovascular Medicine, Hyōgo
  - Tsuchiura Kyodo General Hospital_Internal Medicine, Ibaraki
  - Mito Saiseikai General Hospital_Cardiology, Ibaraki
  - Ishikawa Prefectural Central Hospital_Cardiology, Ishikawa
  - Kanto Rosai Hospital_Cardiology, Kanagawa
  - Yokohama Municipal Citizen's Hospital_Cardiology, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital_Cardiology, Kanagawa
  - Yokohama City University Medical Center_Cardiovascular Center, Kanagawa
  - Yokohama City University Hospital, Kanagawa
  - Tokai University Hospital_Cardiology, Kanagawa
  - National Hospital Organization Kumamoto Medical Center_Cardiology, Kumamoto
  - NHO Kure Medical Center and Chugoku Cancer Center, Kure-shi, Hiroshima
  - The Sakakibara Heart Institute of Okayama_Department of Cardiovascular Medicine, Okayama
  - Osaka General Medical Center_Cardiology, Osaka
  - Ishikiriseiki Hospital_Circulatory Medicine, Osaka
  - Tohoku University Hospital, Cardiovascular, Sendai-shi, Miyagi
  - Shiga University of Medical Science Hospital_Cardiology, Shiga
  - Juntendo University Shizuoka Hospital_Gastroenterology & Hepatology, Shizuoka
  - Juntendo University Shizuoka Hospital, Shizuoka
  - Kagawa Prefectural Central Hospital_Cardiovascular Medicine, Takamatsu-shi, Kagawa
  - Tokushima Prefectural Central Hospital_Cardiology, Tokushima
  - Teikyo University Hospital_Cardiology, Tokyo
  - Tsukuba Medical Center Hospital_Department of Cardiology, Tsukuba-shi, Ibaraki
  - Saiseikai Yokohamashi Nanbu Hospital_Cardiology, Yokohama-shi, Kanagawa
- Malaysia (16):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Sultan Ahmad Shah Medical Centre @IIUM, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun Ipoh, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Sarawak Heart Centre, Kota Samarahan, Sarawak
  - Hospital Serdang, Kajang, Selangor
  - Universiti Teknologi MARA, Sungai Buloh Campus, Sungai Buloh, Selangor
  - Hospital Universiti Sains Malaysia_Kota Bharu, Kelantan, Kota Bharu, Kelantan
  - National Heart Institute, Kuala Lumpur
  - Hospital Universiti Kebangsaan Malaysia, Kuala Lumpur
  - Hospital Queen Elizabeth II, Sabak Bernam
- Mexico (20):
  - Hospital Cardiológica Aguascalientes, Aguascalientes, Aguascalientes
  - Unidad Medica de Alta Especialidad No. 71 IMSS, Torreón, Coahuila
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Nuevo Hospital Civil "Dr. Juan I. Menchaca", Guadalajara, Jalisco
  - Centro de Imagen y Tecnologia en Intervención Cardiovascular, México, La Magdalena Contreras
  - Instituto Nacional de Ciencias Médicas y Nutrición, Tlalpan, Mexico City
  - Hospital General de México (HGM), Cuauhtémoc, México, D.F.
  - UMAE Hospital IMSS, Monterrey, Nuevo León
  - Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León
  - Hospital Angeles de Culiacan, Culiacán, Sinaloa
  - Hermosillo Heart Team, Hermosillo, Sonora
  - Hospital Angeles de las Lomas, México, State of Mexico
  - Hospital Angeles de Xalapa, Xalapa, Veracruz
  - Hospital Juárez de Mexico, Ciudad de México, D.F.
  - Centro Médico Nacional Siglo XXI, Mexico City
  - Instituto Nacional de Cardiología Ignacio Chávez, Mexico City
  - Centro de Estudios Clinicos de Querétaro S.C., Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosi (CICAP), San Luis Potosí City
  - Centro de Atención e Investigación Cardiovascular del Potosi, San Luis Potosí City
  - Servicios Integrales Nova de Monterrey, San Nicolás de los Garza
- Netherlands (18):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - OLVG Oost, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Groene Hart Ziekenhuis, locatie Bleuland, Gouda
  - UMC Groningen, Groningen
  - Tergooi, locatie Hilversum, Hilversum
  - Radboudumc, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Bravis Ziekenhuis, Roosendaal
  - Maasstad Ziekenhuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Medisch Centrum Haaglanden Locatie Westeinde Ziekenhuis, The Hague
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
- Poland (50):
  - Zespol Zakladow Opieki Zdrowotnej w Ostrowie Wielkopolskim, Ostrów Wielkopolski, Greater Poland Voivodeship
  - Zespół Zakładów Opieki Zdrowotnej w Ostrowie Wielkopolskim, Ostrów Wielkopolski, Greater Poland Voivodeship
  - American Heart of Poland S.A., Chrzanów, Lesser Poland Voivodeship
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej We Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej W Pulawach, Puławy, Lublin Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych i Administracji w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - Szpitale Pomorskie Sp. z o.o., Gdynia, Pomeranian Voivodeship
  - American Heart of Poland S.A., Dąbrowa Górnicza, Silesian Voivodeship
  - Szpital Miejski Nr 4 w Gliwicach Sp. z o.o., Oddzial Kardiologii, Gliwice, Silesian Voivodeship
  - American Heart of Poland S.A., Tychy, Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Wojewodzki Szpital Specjalistyczny W Bialej Podlaskiej, Biała Podlaska
  - American Heart of Poland S.A., Bielsko-Biala
  - Szpital Uniwersytecki Nr 2 im. Dr. Jana Biziela, Bydgoszcz
  - 10 Wojskowy Szpital Kliniczny z Polikliniką - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Bydgoszczy, Bydgoszcz
  - Wojewódzki Szpital Specjalistyczny im. NMP w Częstochowie, Częstochowa
  - SCANMED Spółka Akcyjna, Częstochowa
  - Wojewodzki Szpital Zespolony W Elblagu samodzielny publiczny zakład opieki zdrowotnej, Elblag
  - Uniwersyteckie Centrum Kliniczne (UCK), Gdansk
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni Im.Sw.Jana Pawla II, Grodzisk Mazowiecki
  - American Heart of Poland S.A., Kędzierzyn-Koźle
  - SCANMED Spółka Akcyjna, Kluczbork
  - Wojewódzki Szpital Zespolony im. dr. Romana Ostrzyckiego w Koninie, Konin
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Intercard Spolka z ograniczona odpowiedzialnoscia, Krosno
  - SCANMED Spółka Akcyjna, Kutno
  - Uniwersytecki Szpital Kliniczny nr 2 Uniwersytetu Medycznego w Łodzi, Lodz
  - Wojewódzki Specjalistyczny Szpital im.Wl. Bieganskiego,, Lodz
  - Miedziowe Centrum Zdrowia s.a., Lubin
  - 1 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Lublin
  - Podhalanski Szpital Specjalistyczny, Nowy Targ
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Samodzielny Publiczny Zespół Zakładów Opieki Zdrowotnej w Ostrowi Mazowieckiej, Ostrów Mazowiecka
  - Intercard Spolka z Ograniczona Odpowiedzialnoscia, Pińczów
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan
  - Wojewodzki Szpital Im. Sw.Ojca Pio W Przemyslu, Przemyśl
  - Samodzielny Publiczny Zespol Opieki Zdrowotnej w Swidnicy, Swidnica
  - Uniwersytecki Szpital Kliniczny Nr 2 PUM W Szczecinie, Szczecin
  - Specjalistyczny Szpital Im. E. Szczeklika W Tarnowie, Tarnów
  - Specjalistyczny Szpital Miejski im. M.Kopernika w Toruniu, Torun
  - Śródmiejskie Centrum Kliniczne,II Oddział Kardiologii MSB, Klinika Chorób Serca CMKP, Warsaw
  - Szpital Wolski im. dr Anny Gostyńskiej Sp. z o.o., Warsaw
  - Uniwersyteckie Centrum Kliniczne WUM, Warsaw
  - Szpital Grochowski im. dr med. Rafała Masztaka Sp. z o.o., Warsaw
  - Narodowy Instytut Kardiologii Stefana Kardynala Wyszynskiego Panstwowy Instytut Badawczy, Warsaw
  - Wojewodzki Szpital Specjalistyczny We Wroclawiu, Wroclaw
  - Dolnoslaski Szpital Specjalistyczny Im. T.Marciniaka-Centrum Medycyny Ratunkowej, Wroclaw
  - American Heart Of Poland S.A., Zgierz
- South Korea (26):
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - MyongJi Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Inje University Haeundae Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Wonju Severance Christian Hospital, Gangwon-do
  - Chonnam National University Hospital, Gwangju
  - Ajou University Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chungnam National University Sejong Hospital, Sejong-si
  - Kyunghee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang university seoul hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (23):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Univ. Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario Dr. Balmis, Alicante
  - Bellvitge Universitary Hospital, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de Lleida "Arnau de Vilanova", Lleida
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Virgen de la Victoria, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clinico de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari Joan XXIII, Tarragona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Alvaro Cunqueiro de Vigo, Vigo
- Turkey (Türkiye) (34):
  - Ankara Üniversitesi Tıp Fakültesi İbni Sina Hastanesi- Kardiyoloji, Ankara, Altindag
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul, Bakirkoy
  - İstanbul Üniversitesi Cerrahpaşa Tıp Fakültesi Hastanesi- Prof. Dr. Murat Dilmener Yerleşkesi, Istanbul, Bakirkoy
  - Eskişehir Osmangazi Üniversitesi Hastanesi- Kardiyoloji, Eskişehir, Odunpazari
  - Afyonkarahisar Sağlık Bilimleri Üniversitesi Sağlık Uygulama Ve Araştırma Merkezi- Kardiyoloji, Afyonkarahisar
  - Ankara Bilkent Şehir Hastanesi-Kardiyoloji, Ankara
  - Ankara Sehir Hastanesi Cardiology, Ankara
  - Akdeniz Üniversitesi Hastanesi-Kardiyoloji, Antalya
  - Bursa Şehir Hastanesi- Kardiyoloji, Bursa
  - Bursa Yüksek İhtisas Eğitim ve Araştırma Merkezi-Kardiyoloji, Bursa
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Edirne
  - Cerrahpaşa Kardiyoloji Enstitüsü, Istanbul
  - İstanbul Üniversitesi-Cerrahpaşa Tıp Fakültesi Kardiyoloji Enstitüsü, Istanbul
  - Adana Şehir Eğitim ve Araştırma Hastanesi, Istanbul
  - Dr. Siyami Ersek Göğüs Kalp ve Damar Cerrahisi EAH- Kardiyoloji, Istanbul
  - Kartal Kosuyolu Yuksek Ihtisas EAH, Istanbul
  - Koşuyolu Yüksek İhtisas EAH- Kardiyoloji, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Marmara Üniversitesi Pendik EAH- Başıbüyük Yerleşkesi- Kardiyoloji, Istanbul
  - Erciyes University Cardiology, Kayseri
  - Erciyes Üniversitesi Hastanesi- Kardiyoloji, Kayseri
  - Kayseri City Hospital, Kayseri
  - Kayseri Şehir Hastanesi-Kardiyoloji, Kayseri
  - Kocaeli Üniversitesi Hastanesi- Kardiyoloji, Kocaeli
  - Necmettin Erbakan University Hospital, Konya
  - Necmettin Erbakan Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Konya
  - Kütahya Şehir Hastanesi-Kardiyoloji, Kütahya
  - Kütahya Sağlık Bilimleri Üniversitesi Evliya Çelebi EAH- Kardiyoloji, Merkez/Kütahya
  - Mersin Şehir Eğitim Araştırma Hastanesi- Kardiyoloji, Mersin
  - Mersin Üniversitesi Hastanesi- Kardiyoloji, Mersin
  - Antalya Eğitim ve Araştırma Hastanesi- Kardiyoloji, Muratpasa/ Antalya
  - Eskişehir Şehir Hastanesi- Kardiyoloji, Odunpazarı /Eskişehir
  - Ondokuz Mayıs Üniversitesi Hastanesi- Kardiyoloji, Samsun
  - Tokat Gaziosmanpaşa Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Tokat Province
- United Kingdom (27):
  - Royal Cornwall Hospital (Treliske), Truro, Cornwall
  - Royal Bournemouth Hospital - Cardiology, Bournemouth, Dorset
  - William Harvey Hospital, Ashford, Kent
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Harefield Hospital, Harefield, Middlesex
  - Royal Brompton and Harefield Hospitals, Harefield, Middlesex
  - Royal Infirmary of Edinburgh - Cardiology, Edinburgh
  - Golden Jubilee University National Hospital, Glasgow
  - Kettering General Hospital, Kettering
  - Glenfield Hospital, Leicester
  - Lincoln County Hospital, Lincoln
  - Liverpool Heart & Chest Hospital, Liverpool
  - Barts Heart Centre, London
  - St Bartholomew's Hospital - Barts Heart Centre, London
  - Kings College Hospital - Cardiology, London
  - Kings College Hospital, London
  - The James Cook University Hospital - Cardiology, Middlesbrough
  - Freeman Hospital, Newcastle, Newcastle upon Tyne
  - Derriford Hospital - Plymouth, Plymouth
  - Queen Alexandra Hospital - Cardiology, Portsmouth
  - Queen Alexandra Hospital, Portsmouth
  - Northern General Hospital, Sheffield
  - Lister Hospital, Stevenage
  - Morriston Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - Torbay Hospital, Torquay
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com